CLINICAL TRIAL: NCT06551077
Title: Prospective Trial of Posterior Rectus Sheath Hiatal Augmentation (PORSHA) in Paraesophageal Hernia Repair
Brief Title: Posterior Rectus Sheath Hiatal Augmentation in Paraesophageal Hernia Repair
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB24-0322
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Paraesophageal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: POSTERIOR RECTUS SHEATH HIATAL AUGMENTATION (PORSHA) — Use of a novel permanent autologous vascularized biologic fascial flap to reconstruct the diaphragmatic hiatus following standard hiatal hernia repair in selected patients. This technique is called a posterior rectus sheath flap hiatal augmentation or PoRSHA.

SUMMARY:
This study will be a prospective observation study of the use of PoRSHA for repair in patients with challenging paraesophageal hernias.

One of the most challenging problems facing foregut surgeons is the large and complex paraesophageal hernia (PEH) repair in the older patient. The investigator has demonstrated good outcomes and durability with the initial use of a novel permanent autologous vascularized biologic fascial flap to reconstruct the diaphragmatic hiatus following standard hiatal hernia repair in selected patients. This technique is called a posterior rectus sheath flap hiatal augmentation or PoRSHA, which is performed to enhance the hiatal repair for large (type III and IV) and recurrent PEH. The investigator believes by using the patient's autologous vascularized and peritonealized fascia at the hiatal defect, PoRSHA could increase the strength and restore the hiatal complex properties in ways that synthetic mesh, or a primary repair cannot.

The hypothesis is that PoRSHA is a unique technique that has the potential to supplant current approaches to primary hiatal closure in select cases. By augmenting the hiatal closure with a vascularized fascial sheath, PoRSHA provides the tensile strength needed for the attenuated defects in large and complex PEHs.

DETAILED DESCRIPTION:
One of the most challenging problems facing foregut surgeons is the large and complex paraesophageal hernia (PEH) repair in the older patient. Patients often present for surgery after decades of chronic reflux disease and a known hiatal hernia that has finally progressed to a complete intrathoracic stomach with symptoms concerning for a gastric volvulus. Surgery in such patients involves extensive mediastinal dissection to reduce the large hernia sac, repositioning of the gastroesophageal junction into the abdomen and then repair of a significantly attenuated defect in older patients with attenuated diaphragmatic muscle integrity. Challenges with PEH repair are multifactorial and include primary closure of weakened crural muscle in a large attenuated diaphragmatic defect; the absence of a substantial fascial layer to use to close the defect; and the avoidance of permanent mesh due to the risk of shrinkage, dysphagia and esophageal erosion. While a tension free repair is the goal, the use of relaxing incisions, fixation to posterior structures, and other such modifications have not proven to be universally beneficial.

One of the most challenging problems facing foregut surgeons is the large and complex paraesophageal hernia (PEH) repair in the older patient. The investigator has demonstrated good outcomes and durability with the initial use of a novel permanent autologous vascularized biologic fascial flap to reconstruct the diaphragmatic hiatus following standard hiatal hernia repair in selected patients. This technique is called a posterior rectus sheath flap hiatal augmentation or PoRSHA, which is performed to enhance the hiatal repair for large (type III and IV) and recurrent PEH. The investigator believes by using the patient's autologous vascularized and peritonealized fascia at the hiatal defect, PoRSHA could increase the strength and restore the hiatal complex properties in ways that synthetic mesh, or a primary repair cannot.

While initial use of this technique is promising, the investigator believes that long-term and large patient population is necessary to better evaluate the outcomes. The use of the IDEAL framework (Idea, Development, Exploration, Assessment and Long-term follow-up) framework for surgical innovation, to determine its safe development and overall evaluation as a surgical innovation. Using this framework the investigators will evaluate the long-term outcomes in a large patient population.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing PoRSHA. PoRSHA will be offered to all patients with PEH defects measuring greater than 4 cm.

Exclusion Criteria:

* Patients that did not have PoRSHA.
* Patients requiring therapeutic anticoagulation perioperatively or those with bleeding disorders, considering the added risk of bleeding at the donor site with exposed rectus muscle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent PoRSHA at UCMC. We estimate 80-100 patients per year. This study is for all racial and ethnic origins.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrence of hernia as seen radiographically at routine esophagram | At 6 months, 2 year and 5 years' time points

SECONDARY OUTCOMES:
Number or participants with Symptom Relief | At 6 months, 2 year and 5 years' time points
Number of participants with use of anti-acid medications | At 6 months, 2 year and 5 years' time points
Number of participants with dysphagia symptoms | At 6 months, 2 year and 5 years' time points
Number of participants with abdominal wall deformities or symptoms | At 6 months, 2 year and 5 years' time points

CONTACTS AND LOCATIONS:
Overall Officials: Yalini Vigneswaran, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No